CLINICAL TRIAL: NCT04705727
Title: Comparison of the Efficacy and Safety of Budesonide/Formoterol Turbuhaler® Versus Terbutaline Nebulization as Reliever Therapy in Children With Asthma Presenting at the Emergency Room for Moderate Exacerbation
Brief Title: Budesonide/Formoterol Turbuhaler® Versus Terbutaline Nebulization as Reliever Therapy in Children With Moderate Asthma Exacerbation
Acronym: ASTHMAFAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough recruitment in th trial
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTHMAFAST
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- budesonide/formoterol Turbuhaler® (Experimental): After randomization, patients in the experimental arm will receive budesonide/formoterol Turbuhaler® 100/6 μg, one inhalation every 5 minutes (Maximum 12 inhalations).
  Interventions: Drug: Budesonide Formoterol Drug Combination
- nebulisation of terbutaline (Active Comparator): 0.1 mg/kg nebulized terbutaline 5 mg/2 ml of Terbutaline dilution diluted with 2 ml normal saline delivered by an air compressor nebuliser driven by oxygen at a flow rate of 8l/min. The duration of one dose will be approximately 20 minutes and a total of 3 doses will be administered. In case of an insufficient response, 3 additional doses will be administered for a maximum of 6 nebulisations.
  Interventions: Drug: nebulisation of terbutaline

INTERVENTIONS:
Drug: Budesonide Formoterol Drug Combination — This combination will be used to treat the asthma exacerbation, patients will take one inhalation of budesonide/formoterol Turbuhaler® 100/6 μg every 5 minutes (Maximum 12 inhalations).
  Arms: budesonide/formoterol Turbuhaler®
Drug: nebulisation of terbutaline — Patients will receive 0.1 mg/kg nebulized terbutaline 5 mg/2 ml of Terbutaline dilution diluted with 2 ml normal saline delivered by an air compressor nebuliser driven by oxygen at a flow rate of 8l/min. The duration of one dose will be approximately 20 minutes and a total of 3 doses will be administered.
  Arms: nebulisation of terbutaline

SUMMARY:
Combined use of inhaled corticosteroids and long-acting β-agonists (LABAs) as the controller and the quick relief therapy termed single maintenance and reliever therapy (SMART) is a potential therapeutic regimen for the management of persistent asthma. A recent systematic review supports the combined use of inhaled corticosteroids and LABA as both the controller and quick relief therapy (SMART) among patients aged 12 years. In Emergency room (ER), Meta-analysis showed that using salbutamol (or albuterol) by meter doses inhaler (MDI) with a valved holding chamber (VHC) in children with moderate-severe acute asthma exacerbation was more effective, that is, fewer hospital admissions, more clinical improvement, and had fewer adverse effects (tremor and tachycardia) than salbutamol by nebulizer. Therefore, several international guidelines recommend the use of salbutamol by MDI rather than by nebulizer for moderate-severe asthma exacerbations. In children older than 8 years old, dry-powder inhaler (DPI), a device that delivers medication to the lungs in the form of a dry powder is currently used for maintenance and reliever therapy rather than MDI. In this context, we aim to assess the use of combined inhaled corticosteroids and long-acting β-agonists (LABAs) as a quick relief therapy in children older than 8 years old presenting at the ER with moderate asthma exacerbation. Acute asthma patients who had severe exacerbation were excluded from this study (these patients receiving systematically continuous nebulized salbutamol and/or intravenous salbutamol upon their arrival)

ELIGIBILITY:
Inclusion Criteria:

* Children 8-17 years
* Children consulting to the ER with moderate asthma exacerbation (defined by the Pulmonary Score > 3 and ≤7)
* Score for the inhalation technique = 3
* French social security affiliation

Exclusion Criteria:

* Pneumonia
* Pulmonary and/or cardiac congenital malformations
* Chronic pulmonary disease other than asthma (bronchopulmonary dysplasia, cystic fibrosis, or post infectious bronchiolitis obliterans)
* Foreign body aspiration
* Neurological alteration
* Severe asthma exacerbation defined by Pulmonary Score > 7
* Cardiopulmonary failure imminent or mechanical ventilation indication
* Thyrotoxicosis, pheochromocytoma, type 2 diabetes, untreated hypokalemia, obstructive cardiomyopathy, idiopathic subvalvular aortic stenosis, severe hypertension, aneurysm or other serious cardiovascular disorders such as ischemic heart disease, tachyarrhythmias or severe heart failure.
* Pregnancy
* Breastfeeding woman
* Ongoing participation in RIPH1 Intervention Research
* History of intolerance to terbutaline
* Hypersensitivity to the active ingredient or any excipients of terbutaline
* Hypersensitivity (allergy) to budesonide, formoterol or any component of the product (lactose may contain milk proteins in small quantities)
* Patient with an ongoing treatment of itraconazole, ritonavir or other potent CYP3A4 inhibitor, quinidine, disopyramide, procainamide, phenothiazines, antihistamines (terfenadine), monoamine oxidase inhibitors (MAOIs), beta-blockers (including eyedrops) and tricyclic antidepressants

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Percentage of success | Up 30 minutes after the last administration
  Percentage of success define by a pulmonary score < 3 according to the number of administrations necessary to obtain this score.

SECONDARY OUTCOMES:
Number of hospitalized patients | during the month following the asthma attack
  Number of hospitalized patients
Time spent in ER | Up to discharge from the emergency room
  Number of hours of stay in the ER
Score for the inhalation technique | Immediately after each inhalation procedure
  Score for the inhalation technique at each procedure from 0 to 3
Score on the Asthma Control Questionnaire (ACT) | 1 week after randomisation
  Score on the Asthma Control Questionnaire (ACT)
Score on the Asthma Control Questionnaire (ACT) | 1 month after randomisation
  Score on the Asthma Control Questionnaire (ACT)
Number of medical visit | 1 week and 1 month following the exacerbation
  Number of medical visits at 1 week and 1 month following the exacerbation
controlled asthma | 1 month following the exacerbation
  Number of patients with a controlled asthma at 1 month following the exacerbation
Adverse events | Up to 1 month following the exacerbation
  Number of adverse events
FEV1 | 1 month
  FEV1 volume at 1 month
Total pulmonary capacity | 1 month
  Total pulmonary capacity at 1 month
Vital capacity (VC) | 1 month
  Vital capacity volume at 1 month
FEV1/FVC ratio | 1 month
  FEV1/FVC ratio at 1 month
Pulmonary score | Within 5 minutes following each inhalation procedure
  Pulmonary score at each procedure from 0 to 9
Oxygen saturation | Within 5 minutes following each inhalation procedure
  Oxygen saturation at each procedure expressed as a percentage
Respiratory rate | Within 5 minutes following each inhalation procedure
  Respiratory rate number of breathing cycles per minute

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CHU Antoine Béclère, Clamart
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHI Créteil, Créteil
  - Grand Hôpital de l'Est Francilien, Jossigny
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - CHI Villeneuve-Saint-Georges, Villeneuve-Saint-Georges